CLINICAL TRIAL: NCT05186961
Title: Determining Pediatric Dysphagia Awareness in Caregivers
Brief Title: Determining Dysphagia Awareness in Caregivers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Sena Nur Begen, Principle investigator, Atılım University
Other Study IDs: GO 20/290
Record Dates: First submitted 2021-12-26; First posted 2022-01-11 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Caregiver Awareness About Dysphagia
Keywords: caregiver; awareness; dysphagia; children
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- caregivers: Person who provided primary care for children younger than 18 years with swallowing disorders.

SUMMARY:
Genetic, neuromuscular, gastrointestinal, cardiorespiratory diseases and congenital abnormalities can cause dysphagia in children (1, 2). Various symptoms such as coughing during or after feeding, vomiting, recurrent lung infections, inability to gaining weight, difficulty in oromotor control, nasal regurgitation, and prolonged feeding time can be seen in children whose growth and development are affected due to dysphagia (3).

The primary aim of dysphagia rehabilitation is; gaining a child's age-appropriate nutritional experience by ensuring safe swallowing; supporting growth and development (1). Rehabilitation consists of active or passive oral motor exercises, sensory training, thickened fluids, positioning and their combinations (4, 5). The caregiver is one of the most important partners of the rehabilitation program and should apply feding modifications and positioning for safe swallowing during each feeding. In addition, the exercise approaches recommended by the health personnel should be performed in order to improve the swallowing function at certain times of the day (5).

According to a study in patients with neurologenic caregivers' failure to comply with dysphagia strategies; chest infections, aspiration pneumonia, prolongation of hospital stay, and adverse clinical outcomes resulting in death (6). Therefore, the role of caregivers is very important in the perisistence and success of rehabilitation is great. The level of knowledge and awareness of the caregiver directly affects the rehabilitation effectiveness.

The knowledge and awareness of the caregiver directly affects the effectiveness of rehabilitation, as it is the caregiver who is most interested and spends time with the child. The caregiver, who has knowledge about dysphagia, symptoms and management, will give the necessary importance to rehabilitation and will be more aware of the child's existing condition. Thus, communication with health personnel will be strengthened, effectiveness of rehabilitation will increase. The aim of this study; to determine the level of knowledge of the caregiver about dysphagias and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Persons who provided primary care for children younger than 18 years with dysphagia

Exclusion Criteria:

* Doesn't accept to participate to study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Persons who provided primary care for children younger than 18 years with swallowing disorders will be included in the study.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Determination of Caregiver Awareness: | 1 hour
  In order to determine the awareness of dysphagia in caregivers will be asked 6 questions follows. The caregiver will be rate their own level of knowledge on a scale of 1-10. The physiotherapist who made the evaluation will score the caregiver's knowledge level between 1 and 10 in line with the answers.
  Caregiver Awareness of Swallowing Disorder Symptoms In order to determine the awareness of the caregiver about the symptoms of swallowing disorders, 10 questions will be asked to the caregiver. The participant will answer each question as yes or no. In addition, the physiotherapist who made the assessment will observe the child during normal feeding and will answer the same questions asked to the participant as yes or no. The difference between the scores of the physiotherapist and caregiver will be used to determine the awareness of the caregiver.

SECONDARY OUTCOMES:
Demographic Information about caregiver | 1 hour
  Age, gender, occupation, education level, family status, and duration of care for a child with swallowing disorder will be recorded.
Child's Demographic Information | 1 hour
  The child's age, gender, diagnosis, other accompanying diseases, nutritional status (oral, non-oral) will be recorded.
Evaluation of Dysphagia | 1 hour
  Pediatric Eating Assessment Tool (PEDI-EAT-10) will be used to determine dysphagia severity and risk of aspiration. PEDI-EAT-10 is a questionnaire consisting of 10 questions answered by caregivers. It scores between 0-40, an increase in the score indicates an increase in the severity of swallowing disorder. (7)
Chewing Function: | 1 hour
  Karaduman Chewing Performance Scale (KCPS) developed by developed by Arslan et al., chewing function is classified at 5 different levels between 0 - 4 (Level 0= normal chewing function, Level 4= The child cannot bite and chew)(8).
Drooling: | 1 hour
  Drooling intensity and frequency scale (DSFS) is a valid method used in children. Drooling intensity is examined at 5 levels and drooling frequency is examined at 4 different levels (9).
Tongue Trust: | 1 hour
  The tongue trust rating scale (TTRS), developed by Arslan et al., classifies the tongue thrust reflex severity between 0 and 3 according to the position of the tongue at rest (Level 0= no tongue trust, Level 3= severe tongue trust)(10).

CONTACTS AND LOCATIONS:
Overall Officials: Selen Serel Arslan, assoc. prof., Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation Ankara, TURKEY; Sena Begen, Principal Investigator — Atilim University, Facultyof Health Sciences Department of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No
The data obtained will be collected in Excel and SPSS files only on the computer whose password is known by the researchers.

REFERENCES:
- [Background] Lefton-Greif MA. Pediatric dysphagia. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):837-51, ix. doi: 10.1016/j.pmr.2008.05.007. PMID 18940644
- [Background] Prasse JE, Kikano GE. An overview of pediatric dysphagia. Clin Pediatr (Phila). 2009 Apr;48(3):247-51. doi: 10.1177/0009922808327323. Epub 2008 Nov 20. PMID 19023104
- [Background] van den Engel-Hoek L, Harding C, van Gerven M, Cockerill H. Pediatric feeding and swallowing rehabilitation: An overview. J Pediatr Rehabil Med. 2017 May 16;10(2):95-105. doi: 10.3233/PRM-170435. PMID 28582882
- [Background] Chadwick, D. D., Jolliffe, J., & Goldbart, J. (2003). Dysphagia management for adults with learning disabilities: Caregiver knowledge and barriers to their adherence.
- [Background] Serel Arslan S, Kilinc HE, Yasaroglu OF, Demir N, Karaduman AA. The pediatric version of the eating assessment tool-10 has discriminant ability to detect aspiration in children with neurological impairments. Neurogastroenterol Motil. 2018 Nov;30(11):e13432. doi: 10.1111/nmo.13432. Epub 2018 Aug 13. PMID 30101572
- [Background] Serel Arslan S, Aydin G, Alemdaroglu I, Tunca Yilmaz O, Karaduman AA. Reliability and validity of the Karaduman Chewing Performance Scale in paediatric neuromuscular diseases: A system for classification of chewing disorders. J Oral Rehabil. 2018 Jul;45(7):526-531. doi: 10.1111/joor.12642. Epub 2018 May 20. PMID 29727486
- [Background] Rashnoo P, Daniel SJ. Drooling quantification: Correlation of different techniques. Int J Pediatr Otorhinolaryngol. 2015 Aug;79(8):1201-5. doi: 10.1016/j.ijporl.2015.05.010. Epub 2015 May 18. PMID 26092552
- [Background] Serel Arslan S, Demir N, Karaduman AA. Reliability and validity of a tool to measure the severity of tongue thrust in children: the Tongue Thrust Rating Scale. J Oral Rehabil. 2017 Feb;44(2):119-124. doi: 10.1111/joor.12471. PMID 27973693
- [Result] Borowitz KC, Borowitz SM. Feeding Problems in Infants and Children: Assessment and Etiology. Pediatr Clin North Am. 2018 Feb;65(1):59-72. doi: 10.1016/j.pcl.2017.08.021. PMID 29173720